CLINICAL TRIAL: NCT00763438
Title: A Prospective, Open-label, Single-arm, Multinational, Multi-centre, Flexible-dose, Extension Study of the SCoP 99824 With Sertindole for Patients Suffering From Schizophrenia
Brief Title: Safety Study of an Antipsychotic, Sertindole, to Treat Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12009A; 2007.002160-10 (EudraCT Number); NCT00563550 (obsolete NCT alias)
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Sertindole; Safety study
MeSH Terms: conditions — Schizophrenia | interventions — sertindole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sertindole (Experimental)
  Interventions: Drug: Sertindole

INTERVENTIONS:
Drug: Sertindole — Flexible dose

SUMMARY:
The purpose of this study is to permit the patients with schizophrenia who received Sertindole during a previous randomised trial, study 99824, to continue with this treatment.

DETAILED DESCRIPTION:
Schizophrenia is a disabling and often chronic disorder that may require long-term treatment. This protocol is an extension study of a randomised study comparing the safety of Sertindole versus Risperidone. Patients who were randomised to Sertindole and who completed the previous study have the possibility to receive continued Sertindole treatment in this open one-arm study. Sertindole is generally well tolerated and is approved in the EU, but not yet marketed in France. The follow-up of the patients will be similar to that in the previous study and requires quarterly visits. Patient management reflects routine clinical practice in accordance with the Sertindole label. Any severe safety issue is reported to the company.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the previous SCoP study, 99824
* Still fulfils the EU SPC requirements for Sertindole

Exclusion Criteria:

* Withdrawn before the end of the SCoP study, 99824
* Become homeless
* Participation in another clinical trial at the same time
* Unlikely to comply with the clinical study protocol or is unsuitable for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
All serious adverse events reported; visits scheduled every 3 months | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- FR002, Allonnes, France

REFERENCES:
- Available data/document: EMA EudraCT Results: 2007-002160-10 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2007-002160-10/results